CLINICAL TRIAL: NCT05830708
Title: The Efficacy of Probiotics for the Treatment of Alcohol Use Disorder Among Adult Males: A Comparison With Placebo and Acceptance and Commitment Therapy in a Randomized Controlled Trial
Brief Title: The Efficacy of Probiotics for the Treatment of Alcohol Use Disorder Among Adult Males
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Henan Medical University (Other)
Responsible Party: Principal Investigator, Mohammad Farris Iman Leong Bin Abdullah, Principal investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XYEFYLL-(research)-2022-28
Record Dates: First submitted 2023-03-31; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Alcohol Use Disorder
Keywords: probiotics; acceptance and commitment therapy; alcohol use disorder; alcohol craving
MeSH Terms: conditions — Alcoholism | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Three-armed, parallel-group, single-blind, multi-center randomized control trial
Who Masked: Care Provider, Investigator
Masking Description: The randomization will be performed by the study statistician, who had no contact with the patients and not involve in the research project. The statistician is trained to randomize subjects who first enrol in the study into the three groups using computer system for randomization purpose. The allocation sequence will not be available to any member of the research team until databases had been completed and locked. Data collection will be performed by research assistants who were not involved in the study and do not know the objectives of the study. While data analysis will be carried out by the statisticians not involved in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic group (Experimental): Probiotics + conventional drug therapy: treatment includes conventional drug therapy* (initial 2 weeks), then probiotics powder 2g, mixed into water or milk, dissolved and oral; 1 sachet per day for 12 weeks
  *Conventional drug treatment: alcohol detoxification treatment was carried out at the early stage of admission, mainly with benzodiazepine replacement therapy, while adequate supplementation of B vitamins, strengthening symptomatic supportive treatment, and corresponding antipsychotic drugs, antidepressants or emotional stabilizers were given according to the condition. Benzodiazepines are gradually discontinued after withdrawal symptoms disappear (2 weeks).
  Interventions: Dietary Supplement: Lactobacillus sp. probiotic
- Acceptance and commitment therapy (ACT) group (Active Comparator): ACT + conventional drug therapy: treatment includes conventional drug therapy* (initial 2 weeks), then 50 minutes, once a week ACT session for 8 weeks (8 sessions).
  *Conventional drug treatment: alcohol detoxification treatment was carried out at the early stage of admission, mainly with benzodiazepine replacement therapy, while adequate supplementation of B vitamins, strengthening symptomatic supportive treatment, and corresponding antipsychotic drugs, antidepressants or emotional stabilizers were given according to the condition. Benzodiazepines are gradually discontinued after withdrawal symptoms disappear (2 weeks).
  Interventions: Behavioral: Acceptance and commitment therapy
- Placebo group (Placebo Comparator): Placebo + conventional drug therapy: treatment includes conventional drug therapy* (initial 2 weeks), then maltodextrin of the same weight as the test drug treatment group was mixed into water or milk and orally dissolved; 1 sachet per day for 12 weeks.
  *Conventional drug treatment: alcohol detoxification treatment was carried out at the early stage of admission, mainly with benzodiazepine replacement therapy, while adequate supplementation of B vitamins, strengthening symptomatic supportive treatment, and corresponding antipsychotic drugs, antidepressants or emotional stabilizers were given according to the condition. Benzodiazepines are gradually discontinued after withdrawal symptoms disappear (2 weeks).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus sp. probiotic — The probiotic product contains good bacteria Lactobacillus sp. and primarily maltodextrin as carrier. Sachets of products containing the probiotic appear as light-yellow powder. The probiotic products are kept at storage temperature range below 30oC according to the condition recommended by the manufacturer.
  Arms: Probiotic group
Behavioral: Acceptance and commitment therapy — The ACT session is initiated by building good therapeutic rapport with the subject and gather important information such as experiential avoidance, external barriers, fusion past, unworkable actions, and strength of the subject, followed by formulation of the case. The session may began with coaching subjects on acknowledging and accepting their unpleasant thoughts and feelings. The therapy will also focus on defusion to reduce behavioral avoidance of unpleasant thoughts and feelings by acknowledging them but focus on the values identified. Mindfulness is also practice to allow focus onto the present and surrounding to create awareness among the subjects that they are many things in the surrounding which is more enjoyable that we can enjoy rather than making effort to distract or change or avoid the unpleasant thoughts and feelings.
  Arms: Acceptance and commitment therapy (ACT) group
Dietary Supplement: Placebo — The placebo are in powder form prepare in sachet which is light-yellow in color and should be stored in temperature at below 30oC, which is similar to the appearance of the probiotic. Nevertheless, it contains only maltodextrin in same amount as in the placebo.
  Arms: Placebo group

SUMMARY:
This three-armed, parallel-group, single-blind, multi-center randomized control trial (RCT) aims to evaluate the efficacy of probiotic supplement compared with that of acceptance and commitment therapy (ACT) in ameliorating alcohol craving and severity of alcohol use disorder (AUD) in patients diagnosed with AUD after 2 weeks of in-patient detoxification. In addition, this study also compares the efficacy of probiotic supplement and ACT to mitigate common comorbid of AUD (such as depression and anxiety symptoms); changes in event-related potential (ERP) on electroencephalogram (EEG) monitoring which indicate reduce alcohol craving; and depreciate the serum level of pro-inflammatory cytokines, such as interleukin-1β (IL-1β), interleukin-6 (IL-6), and tumor necrosis factor-α (TNF-α) indicating lowering of systemic inflammation.

In phase I of the study, 120 patients diagnosed with AUD (using Diagnostic and Statistical Manual for Mental Disorders 5th Edition or DSM-5) and 120 healthy controls will be recruited. The measured outcomes to be compared between patients with AUD and healthy non-AUD controls include ERP on EEG monitoring, serum levels of pro-inflammatory cytokines (IL-1β, IL-6, and TNF-α), and the fecal microbiota content. Then, in phase II of the study, 120 AUD patients will be randomized into three groups of intervention in a 1:1:1 ratio (Lactobacillus sp. probiotic, ACT and placebo group; n = 40 per group). The participants in probiotic and placebo groups will then consumed the Lactobacillus sp. Probiotic and placebo 1 sachet once a day of probiotic and placebo, respectively for 12 weeks. While participants in ACT group will undergo training for ACT one session per week for 8 weeks. Outcome assessments will be performed across four time points, such as t0 = before intervention began, t1 = 8 weeks after intervention began, t2 = 12 weeks after intervention began, and t3 = 24 weeks after intervention began. The primary outcomes to be measured are the degree of alcohol craving, alcohol withdrawal, and severity of alcohol use disorder. While the secondary outcomes to be assessed are severity of comorbid depression and anxiety symptoms, serum levels of pro-inflammatory cytokines (IL-1β, IL-6, and TNF-α), changes in ERP on EEG monitoring, and fecal microbiota content.

DETAILED DESCRIPTION:
The study will be conducted in the Second Affiliated Hospital of Xinxiang Medical University (Henan Mental Hospital), Xinxiang, Henan, China and Psychiatric Outpatient Clinic in Advanced Medical and Dental Institute, Universiti Sains Malaysia.

The approval of the study was obtained from the Human Research Ethics Committee of Xinxiang Medical University (code: XYEFYLL-(research)-2022-28) and from the Human Research Ethics Committee of Universiti Sains Malaysia (code: USM/JEPeM/22080546). Prior to participation in the trial, participants will be informed of their right to withdraw from the trial at any time and the data collected will be discarded immediately and will not be used for the study. Participants will be reminded that all personal identifiable information will not be used and only group data will be analyzed and published. They will be assured of their anonymity for participating in the trial. The participants will be assured that the data collected will only be used for research purposes and the findings will not be recorded in their case files. All participants will be assigned a research number for identification purposes, for example "PROB 001". All the data collected from the participants will be stored in the research file which will be locked in a file cabinet, whereby the key will be kept by the principal investigator. Data collected may also be stored in thumb drive and lap top which is only accessible by the research team and the principal investigator.

In order to monitor adverse effect (AE) during the trial, all participants will be given a trial card which contains the name, contact number and email of the members of the research team. They are encouraged to contact the research team member in charge if there is any occurrence of AE. The occurrence of AE will then be reported to the "adverse effect" section of the trial's case report form. The AE which may lead to withdrawal of participants from the trial are: (1) adverse reaction which is not related to the study intervention but cause discomfort to the participants, (2) adverse reaction which is related to the study intervention (probiotic, ACT and/or placebo), and (3) any changes in behavior, temperament, personality, psychotic symptoms, and suicidal tendency that occurred after the study intervention began (probiotic, ACT and/or placebo). All AE should be reported to the Human Research Ethics Committee of Xinxiang Medical University and Universiti Sains Malaysia and investigation should be carried out.

The principal investigator will lead the trial center and will coordinate closely with the research and site coordinators in a day-to-day basis involving in the conduct of the clinical trial, subject recruitment, and data collection. A trial monitoring unit will also be set up which will be chaired by the principal investigator, whereby weekly meeting will be held to discuss on the conduct of the trial, auditing of the trial, and prepare report to be submitted to the Human Ethics Committee of Xinxiang Medical University and Universiti Sains Malaysia. The monitoring of trial data and auditing of the trial will be managed by the clinical trial coordination unit of the 2nd Affiliated Hospital of Xinxiang Medical University and Advanced Medical and Dental Institute, Universiti Sains Malaysia, which are independent of the funder. Interim analysis will be carried out if there is such necessity for premature termination of the trial based on assessment and auditing of the trial data.

Primary objective:

To determine the differences in the severity of alcohol dependence, alcohol withdrawal and craving among patients on Lactobacillus sp., placebo and ACT, at 4 timelines (baseline, 8 weeks after starting intervention, 12 weeks after starting intervention, and 24 weeks after starting intervention which is 12 weeks post termination of intervention).

Secondary objectives:

1. To determine the differences in severity of depression and anxiety symptoms, changes of EEG characteristics, and serum levels of pro-inflammatory cytokines among patients on Lactobacillus sp., placebo and ACT, at 4 timelines (baseline, 8 weeks after starting intervention, 12 weeks after starting intervention, and 24 weeks after starting intervention which is 12 weeks post termination of intervention).
2. To assess the differences in gut microbiota profiles of patients on Lactobacillus sp., placebo and ACT via the use of fecal samples, at 3 timelines (baseline, 2 weeks after starting intervention, and 8 weeks after starting intervention).

In this study, the participants will be recruited from the source population. The source population is all the patients who registered under the 2nd Affiliated Hospital of Xinxiang Medical University (XXMU), China and Outpatient Psychiatry Clinic of Advanced Medical and Dental Institute, Universiti Sains Malaysia with alcohol-related mental illness. Advertisement with posters will be placed on display in the 2nd Affiliated Hospital of XXMU, the Department of Psychiatry, XXMU, and Advanced Medical and Dental Institute, Universiti Sains Malaysia to help in the recruitment of subjects. In this study, patients with alcohol dependence who met the diagnostic criteria of "alcohol use disorder" in DSM-5 were selected as the experimental group. Healthy people who met WHO healthy drinking standards or did not drink were used as the healthy control group. Then, baseline assessment (t0) will commence followed by admission of the experimental group subjects for initial 2 weeks for detoxification (routine treatment). The assessment for experimental group subjects include Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar), Penn Alcohol Craving Scale (PACS), Alcohol Use Disorder Identification Test (AUDIT), Hamilton Depression Rating Scale (HAMD), and Hamilton Anxiety Rating Scale (HAMA) scores, ERP analysis, serum pro-inflammatory cytokine levels, and fecal microbiota analysis. While the assessment for healthy controls include ERP analysis, serum pro-inflammatory cytokine levels, and fecal microbiota analysis. During detoxification, treatment of withdrawal symptoms mainly with benzodiazepine replacement therapy, while adequate supplementation of B vitamins, strengthening symptomatic supportive treatment, and corresponding antipsychotic drugs, antidepressants or emotional stabilizers were given according to the condition. Benzodiazepines are gradually discontinued after withdrawal symptoms resolved. Then, subjects in the experimental group will be randomized into three groups, such as probiotics + routine treatment group, placebo + routine treatment group, and acceptance and commitment therapy (ACT) + routine treatment group. Specific intervention will be administered in the respective groups.

The estimated sample size needed for comparing the fecal microbiota, the serum cytokines, and the EEG and physiological indicators between subjects with alcohol use disorder and healthy controls was computed using the G*Power calculator 3.1.9.7 for calculating mean differences between two independent groups, whereby type I error = 0.05, power = 0.8, allocation ratio = 1:1, and effect size = 0.4 [De Giani et al. (2020)]. The estimated sample size needed was 120 subjects per group (inclusive of 20% of drop out). The estimated sample size needed for the experimental subject was calculated using the G*Power calculator 3.1.9.7 for calculating sample size for repeated measure ANOVA, within-between interaction, wherein type I error = 0.05, power = 0.8, number of groups = 3, number of measurements = 3, effect size = 0.15 [Kazemi et al. (2019)]. The estimated sample size needed was 120 subjects, 40 subjects per group (inclusive of 30% drop out).

A single-blind randomized controlled trial design has been chosen. The eligible AD patients will be randomized 1:1:1 ratio to the three arms of the study according to a computer generated, blocked randomization list. The eligible patients will be assigned to the probiotics group, ACT group, and control group with a treatment code concealed in a closed envelope. The randomization will be performed by the study statistician, who had no contact with the patients and not involve in the research project. The statistician is trained to randomize subjects who first enrol in the study into the three groups using computer system for randomization purpose. The allocation sequence will not be available to any member of the research team until databases had been completed and locked. Data collection will be performed by research assistants who were not involved in the study and do not know the objectives of the study. While data analysis will be carried out by the statisticians not involved in the study. Hence, this study is blinded to the researchers but not blinded for the subjects as the ACT group has no parallel control group.

All data analysis will be performed using SPSS software version 26.0. Descriptive statistics for socio-demographic and clinical characteristics, CIWA-Ar), PACS, AUDIT, HAMD, and HAMA scores, ERP analysis, and serum pro-inflammatory cytokine levels will be computed. All categorical variables will be presented in frequency and percentage, while all continuous variables will be reported in mean and standard deviation or median and interquartile range, depends on normality. Initially, the ERP, fecal microbiota content, and serum levels of pro-inflammatory cytokines (IL-1β, IL-6, and TNF-α) will be compared between the experimental subjects and the healthy controls. The serum levels of pro-inflammatory cytokines (IL-1β, IL-6, and TNF-α) will be compared using independent t-test (if data normally distributed) or Mann-Whitney U test (if data non-normally distributed). The mean difference in the primary outcome (CIWA-Ar, PACS, and AUDIT scores) for the three randomized groups (ACT, probiotic, and palcebo groups) at each specific time point (pre-intervention, 2 weeks at completion of conventional treatment [t0], post-treatment at 8 weeks [t1], post-treatment at 12 weeks [t2], and post-treatment at 24 weeks [t3]) will be assessed using one way analysis of variance (ANOVA) followed by false discovery rate adjustment. For the main pool analysis, mixed ANOVA is used to determine the interaction between the groups (ACT, probiotic, and placebo groups) and time points on the primary outcome; interaction = intervention × time; where time is a within-subject variable and intervention effect is a between-subject variable). The main effects of intervention in the groups and time points will be presented as estimated marginal mean and standard error of mean. The study's primary analysis will follow the intention-to-treat (ITT) principle. The data analysis for the study's secondary outcomes (severity of anxiety and depressive symptoms, pro-inflammatory cytokines, EEG characteristics, and fecal microbiota) will be conducted similarly to the primary outcomes' calculation. Statistical significance will be two-tailed and set to p < 0.05.

To handle any missing data, if the missing data represent less than 5% of the study's total collected data, they will be ignored. If the missing data represent more than 5% but less than 40% of the total collected and are assumed to be randomly missing, then multiple imputation (restricted maximum likelihood estimation) will be performed using Stata 15. However, if the missing data represent more than 40% of the total collected data or are assumed to be missing either not randomly or completely randomly, then only the collected data will be used for the study's analysis, and the missing data will be explained as a research limitation in any publications of the study's findings.

ELIGIBILITY:
Inclusion Criteria (AUD patients):

* Hospitalized patients diagnosed with untreated alcohol use disorder (confirmed by the diagnostic criteria of DSM-5).
* Male, age 18 to 55 years old, Han nationality, junior high school education or above, right-handed.
* Those with normal eyesight, including corrected vision(screened clinically).

Exclusion Criteria (AUD patients):

* The patient suffer from other mental illnesses (screen by DSM-V criteria).
* The patient has allergy reaction to medications use for conventional treatment of alcohol use disorder.
* The patient had a history of organic brain disease, a pacemaker, gastrointestinal surgery, or serious health problems.
* The patient had a history of seizures.
* The patient is complicated with severe physical disease.
* Patient has other drug dependence (except for nicotine dependence).
* The patient took drugs affecting intestinal flora 30 days before and during admission.
* The patient has participated in any other alcohol-related studies or trials within the past 30 days.
* Patients had use any prescription or over-the-counter drugs in the past 30 days that may affect mood or alcohol cravings.

Inclusion Criteria (controls):

* Male, age 18 to 55 years old, Han nationality, junior high school education or above, right-handed.
* No history of psychoactive substance abuse, except tobacco (screen with urine dipstick test).
* Those with normal eyesight, including corrected vision (screen clinically).
* No alcoholic beverages in the last 2 weeks.
* According to the WHO healthy alcohol consumption standard, the average intake of pure alcohol per week is less than 210 grams, or do not drink at all (screen clinically).

Exclusion Criteria (controls):

* Those who suffer from other mental illnesses (screen by DSM-V criteria).
* Those who has history of organic brain disease, a pacemaker, gastrointestinal surgery, or serious health problems.
* Those who has history of seizures.
* Those complicated with severe physical disease.
* Those with drug dependence, including alcohol dependence (exception for nicotine dependence).
* Those who took drugs affecting intestinal flora 30 days before and during admission.
* Those who has participated in any other alcohol-related studies or trials within the past 30 days.
* Those who use any prescription or over-the-counter drugs in the past 30 days that may affect mood or alcohol cravings.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male gender
Enrollment: 120 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Alcohol Use Disorder Identification Test score across four time points | At four time points of assessment: t0 (baseline) = before starting intervention, t1 = 8 weeks after intervention began, t2 = 12 weeks after intervention began, and t3 = 24 weeks after intervention began
  This questionnaire can screen drinkers from mild to severe.The reliability and validity of the Chinese version are 0.782. Factor analysis showed that indeed the Chinese version of the AUDIT comprised of three factors and had good convergent and discriminant validity. The scale consists of 10 questions, of which three relate to the amount and frequency of alcohol consumption, three relate to alcohol dependence and four involve in various problems caused by alcohol. The total score range from 0 to 40. The score of the scale ≥ 8 is positive. In general, those with high scores on the first three questions but low scores on the rest suggest serious harmful drinking; High scores in questions 4, 5 and 6 indicate alcohol dependence; High scores in the final section indicate that drinking has caused harm.
Change in Clinical Institute Withdrawal Assessment for Alcohol-Revised score across four time points | At four time points of assessment: t0 (baseline) = before starting intervention, t1 = 8 weeks after intervention began, t2 = 12 weeks after intervention began, and t3 = 24 weeks after intervention began
  The scale is a standard tool for quantifying the severity of alcohol withdrawal symptoms. The reliability of the Chinese version of CIWA-Ar was good with Cronbach's α of 0.83. The total score range from 0 to 30. The total score < 10 suggests mild withdrawal reaction. The score of 10 to 20 indicates moderate. And the total score of more than 20 is considered severe. A severe total score is associated with a risk of delirium tremens and seizures.
Change in Penn Alcohol Craving Scale score across four time points | At four time points of assessment: t0 (baseline) = before starting intervention, t1 = 8 weeks after intervention began, t2 = 12 weeks after intervention began, and t3 = 24 weeks after intervention began
  This questionnaire consists of five items to evaluate the severity of craving, including frequency, intensity, duration, difficulty of coping, and average craving degree. The reliability of the Chinese version of PACS was good at Cronbach's α of 0.97. Each item is scored in a seven-point Likert scale from 0 to 6, with 0 being none and 6 being extremely severe. Thus, the total score range from 0 to 30. The higher the total score, the greater is the degree of craving. The subjects will be asked to answer questions according to the situation in the past week.

SECONDARY OUTCOMES:
Change in Hamilton Depression Rating Scale score across four time points | At four time points of assessment: t0 (baseline) = before starting intervention, t1 = 8 weeks after intervention began, t2 = 12 weeks after intervention began, and t3 = 24 weeks after intervention began
  The scale is use to assess the emotional aspects of patients.The reliability of the Chinese version of the HAMD was acceptable with Cronbach's α of 0.714. The HAMD we choose is the 24-item version. The total score > 35 indicates severe depression; The total score from 20 to 35 indicates definite depression; And total score from 8 to 20 indicates possible depression. If < 8 points, it is considered normal.
Change in Hamilton Anxiety Rating Scale score across four time points | At four time points of assessment: t0 (baseline) = before starting intervention, t1 = 8 weeks after intervention began, t2 = 12 weeks after intervention began, and t3 = 24 weeks after intervention began
  The scale is use to assess the anxiety symptoms of patients. The reliability of the Chinese version of the HAMA was 0.93. HAMA consists of 14 items. The total score range from 0 to 56. The total score ≥ 29 indicates that there may be serious anxiety; The total score ≥ 21 indicates that there must be obvious anxiety; The total score ≥ 14 indicates that there must be anxiety; And the total score ≥ 7 indicates that there may be anxiety. If < 7 points, it is considered that there are no anxiety symptoms.
Change in event-related potential in EEG monitoring across four time points | At four time points of assessment: t0 (baseline) = before starting intervention, t1 = 8 weeks after intervention began, t2 = 12 weeks after intervention began, and t3 = 24 weeks after intervention began
  Visual stimuli will be presented by E-Prime 2.0 software. The paradigm consists of three types of images such as i) images related to alcohol cues (common drinking environments, habitual drinking products, etc.), ii) neutral images unrelated to alcohol cues, and iii) task-related images requiring key operation. We will collect EEG while patients watch the stimulation paradigm. We will use the Brain Amp MR-32 instrument to collect signals, and record data through the Brian Vision Recorder software. 64 standard scalp positions will be recorded according to the 10-10 standard lead system. The sampling rate is 1000 Hz, and the impedance between electrode and skin should be less than 5 kΩ. EEG monitoring aims to detect and monitor P300. Enhanced P300 response was alcohol-specific and would not be extended to other motivational related stimuli.
Change in serum tumor necrosis factor-α (in ng/mL) across four time points | At four time points of assessment: t0 (baseline) = before starting intervention, t1 = 8 weeks after intervention began, t2 = 12 weeks after intervention began, and t3 = 24 weeks after intervention began
  Serum samples will be analyzed for the interleukins such as interleukin by commercial enzyme-linked immunoabsorbent assay (ELISA) kit following manufacturer's instructions. Samples may need to be diluted with appropriate amounts of buffer provided in the kit to give constant dilutions prior to analyses. A standard curve will be constructed, and the concentration of samples will be read against the standard curve and expressed as concentration per unit of the samples. The modulation of these immunological parameters will also be determined using gene expression analyses using via real-time PCR.
Change in fecal microbiota analysis across three time points | At three time points of assessment: t0 (baseline) = before starting intervention, t1 = 8 weeks after intervention began, and t2 = 12 weeks after intervention began
  Prior to fecal sample collection, an early announcement will be made one or two weeks earlier and all subjects will be given the fecal collection kit. Materials provided for fecal collection, are fecal collection tube (with RNAlater™ solution and 4 glass beads in tube) and rice paper. A piece of rice paper is floated on water surface in a lavatory bowl. Using the spatula attached to the tube cover, two spatula portions of the feces defecated on the rice paper are collected. Fecal specimens should not be contaminated with water, urine, barium, or mineral oil. Spatula is put back into the fecal collection tube and capped tightly. Then put into ziplock bag, sealed, stored in -80℃ (if possible, can be quick-frozen liquid nitrogen). Fecal sample collection must be completed within one week, upon receiving the fecal collection tube and rice paper. A picture instruction leaflet will be provided prior to fecal collection.
Change in serum interleukin-1β (in ng/mL) across across four time points | At four time points of assessment: t0 (baseline) = before starting intervention, t1 = 8 weeks after intervention began, t2 = 12 weeks after intervention began, and t3 = 24 weeks after intervention began
  Serum samples will be analyzed for the interleukins such as interleukin by commercial enzyme-linked immunoabsorbent assay (ELISA) kit following manufacturer's instructions. Samples may need to be diluted with appropriate amounts of buffer provided in the kit to give constant dilutions prior to analyses. A standard curve will be constructed, and the concentration of samples will be read against the standard curve and expressed as concentration per unit of the samples. The modulation of these immunological parameters will also be determined using gene expression analyses using via real-time PCR.
Change in serum interleukin-6 (in ng/mL) across four time points | At four time points of assessment: t0 (baseline) = before starting intervention, t1 = 8 weeks after intervention began, t2 = 12 weeks after intervention began, and t3 = 24 weeks after intervention began
  Serum samples will be analyzed for the interleukins such as interleukin by commercial enzyme-linked immunoabsorbent assay (ELISA) kit following manufacturer's instructions. Samples may need to be diluted with appropriate amounts of buffer provided in the kit to give constant dilutions prior to analyses. A standard curve will be constructed, and the concentration of samples will be read against the standard curve and expressed as concentration per unit of the samples. The modulation of these immunological parameters will also be determined using gene expression analyses using via real-time PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Farris Iman Leong Bin Abdullah, Dr Psych, Principal Investigator — Advanced Medical and Dental Institute, Universiti Sains Malaysia (USM)

REFERENCES:
- [Derived] Zhang B, Zhang R, Deng H, Cui P, Li C, Yang F, Leong Bin Abdullah MFI. Research protocol of the efficacy of probiotics for the treatment of alcohol use disorder among adult males: A comparison with placebo and acceptance and commitment therapy in a randomized controlled trial. PLoS One. 2023 Dec 5;18(12):e0294768. doi: 10.1371/journal.pone.0294768. eCollection 2023. PMID 38051740